CLINICAL TRIAL: NCT03053713
Title: The Effect of Diet Modification on Clinical Disease Activity, the Gut Microbiome and Immune Responses in Patients With Ulcerative Colitis
Brief Title: The Effect of Diet on Disease Activity and Symptoms in Patients With Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, Deanna Gibson, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-03300
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
Keywords: Mediterranean diet pattern; nutrition; diet intervention; disease activity; intestinal microbiome; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Using a randomized, parallel treatment design, the effects of the Mediterranean diet pattern on symptoms, clinical disease activity, gut microbiome and fecal biomarkers in stable UC patients in remission will be examined. Using this design, we will compare the habitual diet (taken as a "control" diet) to the Mediterranean diet pattern taken by UC patients over a 12-week period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet Pattern (Active Comparator): Mediterranean diet pattern x 12 weeks.
  Interventions: Behavioral: Mediterranean diet pattern
- Habitual Diet (Placebo Comparator): Habitual diet (control) x 12 weeks.
  Interventions: Behavioral: Habitual diet (control)

INTERVENTIONS:
Behavioral: Mediterranean diet pattern — Subjects assigned to the Mediterranean diet pattern arm will receive nutrition advice from a Registered Dietitian (RD). The RD will meet with the subjects (in-person) to provide diet education at randomization, week 3 and week 6 of the intervention. Phone and e-mail follow-up will occur at week 2 and week 9 to provide cooking tips, recipes, videos and answer questions.
  Arms: Mediterranean Diet Pattern
Behavioral: Habitual diet (control) — Subjects assigned to follow their habitual group will be instructed to make no changes to their diet over 12 weeks.
  Arms: Habitual Diet

SUMMARY:
The Mediterranean Diet Pattern (MDP) has been shown to have beneficial effects on the intestinal bacteria and the immune system in diseases like cancer and diabetes. The aim of this study is to determine if a MDP will have an impact on symptoms, intestinal bacteria and the immune system in Ulcerative Colitis (UC). Symptoms, blood and stool will be examined to determine if the MDP results in changes to the intestinal bacteria or immune system.

DETAILED DESCRIPTION:
Few studies have found a single dietary factor as being protective or detrimental against inflammatory bowel disease (IBD), therefore novel diet approaches for the prevention and treatment of IBD are urgently needed. The Mediterranean Diet Pattern (MDP) is associated with improvements in health status and inflammatory markers in healthy individuals and rodent models of colitis. Reductions in inflammatory biomarkers and a "normalization" of the gut microbiota have been shown in patients with Crohn's disease following a MDP. To date, no studies have examined the effect of MDP on disease activity, inflammatory markers or the effects on the microbiome in ulcerative colitis (UC).

This study will examine the effects of a MDP taken by patients with UC on 1) symptoms, clinical and quality of life endpoints and 2) on gut microbiome and fecal immune biomarkers. One hundred subjects and two subjects with UC will be randomly allocated to follow a MDP for 12 weeks or their usual diet (controls). Upon initiation, throughout and completion of each diet, symptoms, clinical and quality of life endpoints will be monitored. Fecal samples will be collected to assess pH, short-chain fatty acid concentrations, bacterial abundance and diversity.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative Colitis in clinical remission (partial Mayo score 0-1)
* Taking oral 5-ASA, methotrexate, azathioprine or 6-mecaptopurine as long as there have been no changes in dosage for 2 months prior to the start of the study
* Generally healthy besides having UC
* Agree not to use any dietary supplements, herbal treatments, prebiotics, probiotics or diet therapies within three weeks of the onset of the trial or during the study

Exclusion Criteria:

* Using prednisone (or steroid equivalent) or biologics (i.e., infliximab, adalimumab, vedolizumab) at the time of enrollment
* Using antibiotics two weeks prior to or anytime during the study period
* Pregnancy, lactation or desire to become pregnant during the study period because we do not know if or how an unborn baby/fetus could be harmed
* History of colectomy or extensive colonic resection or disease is limited to the rectum
* Significant chronic disorders such as severe cardiac disease, significant renal failure, severe pulmonary disease (need for oxygen)
* Active gastrointestinal infection (e.g., C. difficile infection)
* Severe psychiatric disorder
* Unable or unwilling to consent
* Unable to comply with study requirements
* Presence of alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Simple Clinical Colitis Activity Index (SCCAI) | Change from baseline to week 12
  The SCCAI is a symptom-based disease activity index that uses six clinical parameters: daytime and nocturnal bowel frequency, urgency, amount of blood in the stool, well-being and extraintestinal manifestations. A reduction of SCCAI >1.5 is considered clinically significant and SCCAI score of <4 is indicative of remission.

SECONDARY OUTCOMES:
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | 12 weeks
  Quality of life improvement measured at baseline, week 3, week 6, week 9 and 12.
Fecal microbiota | 12 weeks
  Fecal microbiota measured by examining microbial taxa from stool at baseline and 12 weeks
Change in mucosal inflammation measured by fecal calprotectin | 12 weeks
  Change in mucosal inflammation will be measured by fecal calprotectin at baseline and week 12
Change in serum marker of inflammation (serum CRP) | 12 weeks
  Change in markers of inflammation will be measured by serum CRP
Change in serum marker of inflammation (serum ferritin) | 12 weeks
  Change in markers of inflammation will be measured by serum ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Gibson, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (1):
- University of British Columbia - Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeCoffe D, Quin C, Gill SK, Tasnim N, Brown K, Godovannyi A, Dai C, Abulizi N, Chan YK, Ghosh S, Gibson DL. Dietary Lipid Type, Rather Than Total Number of Calories, Alters Outcomes of Enteric Infection in Mice. J Infect Dis. 2016 Jun 1;213(11):1846-56. doi: 10.1093/infdis/jiw084. Epub 2016 Apr 10. PMID 27067195
- [Background] Strisciuglio C, Giugliano F, Martinelli M, Cenni S, Greco L, Staiano A, Miele E. Impact of Environmental and Familial Factors in a Cohort of Pediatric Patients With Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):569-574. doi: 10.1097/MPG.0000000000001297. PMID 27306105
- [Background] Marlow G, Ellett S, Ferguson IR, Zhu S, Karunasinghe N, Jesuthasan AC, Han DY, Fraser AG, Ferguson LR. Transcriptomics to study the effect of a Mediterranean-inspired diet on inflammation in Crohn's disease patients. Hum Genomics. 2013 Nov 27;7(1):24. doi: 10.1186/1479-7364-7-24. PMID 24283712
- [Derived] Haskey N, Ye J, Josephson J, Raman M, Ghosh S, Gibson DL. Metabolomic Signatures Highlight Fiber-Degrading Bacteroides Species in Mediterranean Diet Response Among Ulcerative Colitis. Gastro Hep Adv. 2024 Dec 31;4(4):100606. doi: 10.1016/j.gastha.2024.100606. eCollection 2025. PMID 40242173
- [Derived] Haskey N, Shim RCK, Davidson-Hunt A, Ye J, Singh S, Dieleman LA, Jacobson K, Ghosh S, Gibson DL. Dietary adherence to the Mediterranean diet pattern in a randomized clinical trial of patients with quiescent ulcerative colitis. Front Nutr. 2022 Dec 21;9:1080156. doi: 10.3389/fnut.2022.1080156. eCollection 2022. PMID 36618690